CLINICAL TRIAL: NCT07019883
Title: A Phase 1 Study to Evaluate the Safety and Immunogenicity of Two Doses of a Novel H5 Antigenically Central (AC)-Anhui mRNA-LNP Vaccine in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Two Doses of a Novel H5 Central Antigen mRNA-LNP in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 24-0024
Record Dates: First submitted 2025-05-29; First posted 2025-06-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09-10

CONDITIONS: Avian Influenza
Keywords: H5N1; Healthy Adults; Influenza; Novel H5 Central Antigen mRNA-LNP; Phase 1; Safety and Immunogenicity; Vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Stage 2 is double-blinded, only individuals delegated to unblinded activities will know study vaccination assignments. As there is no placebo, we do not anticipate unintentional unblinding due to effects of the investigational agents. As the products are physically indistinguishable, no blinding sleeve or unblinded administrator will be required.
  Laboratory personnel performing assays will receive study samples blinded to participant data, as appropriate to avoid introducing bias in immunogenicity analysis.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Stage 1 Group 1 (Experimental): Healthy male and non-pregnant female participants, ages 18 to 49, will be administered two intramuscular doses of H5 Antigenically Central (AC)-Anhui RNA Vaccine at 12.5 mcg on days 1 and 29. N=10
  Interventions: Biological: H5 AC-Anhui RNA Vaccine; Other: Sodium Chloride, 0.9%
- Stage 1 Group 2 (Experimental): Healthy male and non-pregnant female participants, ages 18 to 49, will be administered two intramuscular doses of H5 AC-Anhui RNA Vaccine at 25 mcg on days 1 and 29. N=10
  Interventions: Biological: H5 AC-Anhui RNA Vaccine; Other: Sodium Chloride, 0.9%
- Stage 1 Group 3 (Experimental): After the Protocol Safety Review Team (PSRT) reviews the reactogenicity and safety data, through Day 8, for both Stage 1 Group 1 and Stage 1 Group 2, healthy male and non-pregnant female participants, ages 18 to 49, will be administered two intramuscular doses of H5 AC-Anhui RNA Vaccine at 50 mcg on days 1 and 29. N=10
  Interventions: Biological: H5 AC-Anhui RNA Vaccine; Other: Sodium Chloride, 0.9%
- Stage 2 Group 4 (Experimental): Following the Day 36 Stage 1 Group 3 data review by the Protocol Safety Review Team (PSRT), healthy male and non-pregnant female participants, ages 18 to 49, will be administered two intramuscular doses of H5 AC-Anhui RNA Vaccine at 25 mcg on days 1 and 29. N=25
  Interventions: Biological: H5 AC-Anhui RNA Vaccine; Other: Sodium Chloride, 0.9%
- Stage 2 Group 5 (Experimental): Following the Day 36 Stage 1 Group 3 data review by the Protocol Safety Review Team (PSRT), healthy male and non-pregnant female participants, ages 18 to 49, will be administered two intramuscular doses of H5 Astrakhan RNA Vaccine at 25 mcg on days 1 and 29. N=25
  Interventions: Biological: H5 Astrakhan RNA Vaccine; Other: Sodium Chloride, 0.9%

INTERVENTIONS:
Biological: H5 AC-Anhui RNA Vaccine — A nucleoside-modified mRNA vaccine encoding a stabilized, antigenically central hemagglutinin (HA) from influenza A(H5), based on A/Anhui/1/2005 (clade 2.3.4) with substitutions 222QL, 224GS, 156TA, and 134TA. The 2119-nt mRNA is encapsulated in lipid nanoparticles (LNPs) for intramuscular delivery.
  Arms: Stage 1 Group 1; Stage 1 Group 2; Stage 1 Group 3; Stage 2 Group 4
Biological: H5 Astrakhan RNA Vaccine — The vaccine product consists of a monovalent nucleoside-modified mRNA that encodes a traditionally selected avian influenza HA. The H5 Astrakhan RNA encodes the HA from the clade 2.3.4.4b A/Astrakhan/3212/2020 virus.
  Arms: Stage 2 Group 5
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection

SUMMARY:
This is a phase 1, multicenter, randomized, double-blind trial of two influenza A/H5 mRNA-based vaccines on healthy adult participants, 18-49 years of age. Stage 1 will serve as the open-label, dose finding stage. The first 10 participants will receive 12.5 mcg of H5 AC-Anhui RNA vaccine (Group 1), and the second 10 participants will receive 25 mcg of H5 AC-Anhui RNA vaccine (Group 2). After Protocol Safety Review Team (PSRT) review of reactogenicity and safety data through Day 8 for both Groups 1 and 2, another 10 participants may be enrolled to receive 50 mcg of H5 AC-Anhui RNA vaccine (Group 3). Safety data from 7 days after dose 2 for Groups 1 and 2 participants will be reviewed by the PSRT prior to clearing Group 3 participants for the second dose of vaccine. Individual participants will be followed for approximately 6 months following the second dose of vaccine. The primary objective is to assess the safety of two doses of H5 AC-Anhui RNA vaccine or H5-Astrakhan RNA vaccine administered intramuscularly in healthy adults (18-49 years). Once the Day 36 data from Group 3 are reviewed by the PSRT, a dose will be chosen (12.5 mcg, 25 mcg, or 50 mcg) for advancement to Stage 2 where 50 participants will be randomized 1:1 to receive either H5 AC-Anhui RNA (Group 4) or H5 Astrakhan RNA (Group 5) in a double-blinded manner.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind trial of two influenza A/H5 mRNA-based vaccines. The trial population consists of healthy adult participants, 18-49 years of age. Stage 1 will serve as the open-label, dose finding stage. The first 10 participants will receive 12.5 mcg of H5 AC-Anhui RNA vaccine (Group 1), and the second 10 participants will receive 25 mcg of H5 AC-Anhui RNA vaccine (Group 2). These groups will be enrolled sequentially without pause unless study halting rules are triggered. After Protocol Safety Review Team (PSRT) review of reactogenicity and safety data through Day 8 for both Groups 1 and 2, another 10 participants may be enrolled to receive 50 mcg of H5 AC-Anhui RNA vaccine (Group 3). Safety data from Day 36 (7 days after dose 2) for Groups 1 and 2 participants will be reviewed by the PSRT prior to clearing Group 3 participants for the second dose of vaccine. Once the Day 36 data from Group 3 are reviewed by the PSRT, a dose will be chosen (12.5 mcg, 25 mcg, or 50 mcg) for advancement to Stage 2 where 50 participants will be randomized 1:1 to receive either H5 AC-Anhui RNA (Group 4) or H5 Astrakhan RNA (Group 5) in a double-blinded manner. Participants will be randomized on the day of enrollment. Screening and enrollment can occur on the same day. Individual participants will be followed for approximately 6 months following the second dose of vaccine.

The primary objective is to assess the safety of two doses of H5 AC-Anhui RNA vaccine or H5-Astrakhan RNA vaccine administered intramuscularly in healthy adults (18-49 years). The secondary objective is to assess the serum antibody responses to H5 AC-Anhui RNA vaccine or H5-Astrakhan RNA vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to the initiation of any trial procedures
2. Can understand and agrees to comply with all planned trial procedures and be available for all study visits
3. Adult volunteers, age 18-49 years, inclusive, at time of enrollment.
4. In good general health.* * Good health is defined by the absence of a medical condition described in the exclusion criteria. If the participant has another current, ongoing medical condition, the condition cannot meet any of the following criteria:

   1. was first diagnosed within 3 months of enrollment with a clinically significant condition, in the opinion of investigator
   2. had non-elective surgery, clinically significant medical procedure, or hospitalization within 3 months of enrollment;
   3. received new prescription for systemic medication within 30 days of enrollment, unless the new prescription is in the same class of agent or a transition from generic to/from brand name equivalent; or
   4. takes medication that may pose a risk to participant's safety or impede assessment of adverse events or study endpoints if they participate in the study.
5. Participants of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception.*** *These criteria apply to females who are in a heterosexual relationship who are of childbearing potential. Participants not of childbearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or permanently implanted contraceptive device placement).

   **True abstinence is complete lack of penile-vaginal intercourse. Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods.

   ***Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the participant's vaccination; intrauterine devices; birth control pills; and injectable/implantable/insertable/transdermal hormonal birth control products. Participants must have used >/=1 acceptable primary form of contraception for at least 30 days prior to vaccination and agree to continue >/=1 acceptable primary form of contraception through 60 days after last vaccination.
6. Must agree to refrain from donating blood or blood products during the first 6 months of the study
7. Body mass index (BMI) 18 kg/m^2 to 35 kg/m^2, inclusive, and a weight of 130 kg or less at the time of screening

Exclusion Criteria:

1. Positive pregnancy test at screening or prior to vaccine dose
2. Participant who is lactating
3. Presence of a significant psychiatric condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation
4. History of drug abuse or alcohol abuse within 6 months of enrollment that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation
5. Has a significant acute illness (with or without fever), as determined by the site PI or appropriate sub-investigator, within 72 hours prior to dosing* *If the participant meets all other eligibility criteria, they may be enrolled and dosed once they meet this eligibility criterion. If the illness resolves within the 28-day screening window, they do not need to be rescreened, otherwise they will need to be rescreened
6. Currently enrolled in or plans to participate in another clinical trial with an investigational agent
7. Has a history of anaphylaxis to any drug compound, vaccine, food, or other substance, unless approved by the Investigator (or designee)**

   **Sensitivity to components of the study product is exclusionary.
8. Received any live-attenuated or mRNA vaccine in the 28 days prior or any other vaccine in the 14 days prior to study vaccination
9. Has used any prohibited medication within 30 days prior to Day 1 or plans to use prohibited medications*** through Day 57

   ***Prohibited medications include systemic immunosuppressive drugs, immune modulators (except acetaminophen or non-steroidal anti-inflammatory drugs), oral corticosteroids, and systemic antineoplastic agents. Topical, inhaled, and intranasal steroids, as well as topical anti-neoplastic agents are acceptable
10. Abnormal blood pressure or temperature (Grade 1 or higher) at time of vaccination

    ****Grade 1 or higher is equivalent to: Systolic blood pressure (SBP) > 140 mmHg or < 90 mmHg Diastolic blood pressure (DBP) > 90 mmHg Oral temperature >/= 38.0 degrees Celsius (100.4 degrees Fahrenheit)
11. Abnormal heart rate (Grade 2 or higher) at time of vaccination
12. Known and current human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection, based on medical history
13. Extended exposure (e.g., occupational or home exposure) to cattle or poultry since March 1, 2024
14. Ingestion of non-pasteurized milk since March 1, 2024, or plans to drink non-pasteurized milk during participation in the trial
15. Prior receipt of an influenza A/H5 vaccine
16. History of myocarditis or pericarditis
17. Has any medical disease or condition***** that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation****** *****Medical conditions include, but are not limited to, kidney disease with creatinine clearance < 89 mL/min/1.73 cm2 Chronic Kidney Disease Epidemiology Collaboration method (CKD-EPI); known active liver disease; ischemic heart disease, clinically significant cardiac conduction disorder, arrythmia requiring treatment, congenital long QT syndrome, uncompensated heart failure; diabetes requiring insulin; neuropathy or myopathy; history of Guillain-Barré Syndrome; and malignancy (not including squamous cell skin cancer, basal cell skin cancer, or cervical lowgrade squamous intraepithelial lesions) ******Participation may be precluded due to safety concern or inability to adequately evaluate clinical trial endpoints.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Number and Percentage of participants experiencing any adverse events of special interest (AESI) | Through 90 days after second vaccination
Number and Percentage of participants experiencing any medically attended adverse events (MAAE) | Through 6 months following the second dose
Number and Percentage of participants experiencing any non-serious unsolicited adverse events (AEs) | Through 28 days following each dose
Number and Percentage of participants experiencing any serious adverse events (SAE) | Through 6 months following the second dose
Number and Percentage of participants experiencing new-onset chronic medical conditions (NOCMC) | Through 6 months following the second dose
Number and Percentage of participants experiencing solicited local reactogenicity adverse events (AEs) | Through 7 days following each dose
Number and Percentage of participants experiencing solicited systemic reactogenicity adverse events (AEs) | Through 7 days following each dose
Number and Percentage of participants with clinical laboratory adverse events (AEs) | Through 7 days following each dose

SECONDARY OUTCOMES:
Geometric mean fold rise (GMFR) in Group 1-specific anti-stalk serum antibodies since pre-vaccination (Day 1) | Day 8 through Day 57
Geometric mean fold rise (GMFR) in homologous and heterologous H5-specific Neut antibody since pre-vaccination (Day 1) | Day 8 through Day 57
Geometric mean fold rise in homologous and heterologous H5-specific Hemagglutination Inhibition Antibody (HAI) antibody since pre-vaccination | Day 8 through Day 57
Geometric mean titers of Group 1-specific anti-stalk serum antibodies | Day 1 through Day 57
Geometric mean titers of homologous and heterologous H5-specific hemagglutinin inhibition (HAI) antibodies | Day 1 through Day 57
Geometric mean titers of homologous and heterologous H5-specific neutralizing antibodies (Neut) | Day 1 through Day 57
Number and Percentage of participants achieving Hemagglutination Inhibition Antibody (HAI) titer seroconversion since pre-vaccination (Day 1) against the homologous and heterologous H5-specific hemagglutinin | Day 8 through Day 57
  Seroconversion is defined as either a pre-vaccination titer <1:10 and a post-vaccination titer >/=1:40 or a pre- vaccination titer >/=1:10 and a minimum four-fold rise in post-vaccination antibody titer
Number and Percentage of participants demonstrating Hemagglutination Inhibition Antibody (HAI) titer seroprotection against homologous and heterologous H5-specific hemagglutinin | Day 1 through Day 57
  Seroprotection defined as >/=1:40 titer
The number and percentage of participants achieving Neut seroconversion since pre-vaccination (Day 1) against the homologous and heterologous H5-specific hemagglutinin | Day 8 through Day 57
  Seroconversion is defined as either a pre-vaccination titer <1:10 and a post-vaccination titer >/= 1:40 or a pre-vaccination titer >/= 1:10 and a minimum four-fold rise in post-vaccination antibody titer

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT07019883/ICF_000.pdf